CLINICAL TRIAL: NCT06227182
Title: Ultrasound and Magnetic Resonance Imaging for Assessing Muscle Contractile Performance in FSHD - An Exploratory Study
Brief Title: Magnetic Resonance Imaging and Ultrasound Comparison With Load Evaluation
Acronym: MUSCLE+
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Solve FSHD (Unknown)
Responsible Party: Sponsor
Other Study IDs: NL84168.091.23
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-01

CONDITIONS: Muscular Dystrophy, Facioscapulohumeral
Keywords: Magnetic Resonance Imaging; Muscle Ultrasound
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral | interventions — Electromyography; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy individuals: Healthy individuals between 18 and 70 years old.
  Interventions: Diagnostic Test: Muscle ultrasound with surface electromyography and dynamometry; Diagnostic Test: MRI scan
- Patients with FSHD: Individuals with clinically and genetically proven FSHD type 1 or type 2.
  Interventions: Diagnostic Test: Muscle ultrasound with surface electromyography and dynamometry; Diagnostic Test: MRI scan

INTERVENTIONS:
Diagnostic Test: Muscle ultrasound with surface electromyography and dynamometry — The three procedures are conducted simultaneously for upper and lower extremity muscles. A standard muscle ultrasound preset with a fixed depth of 4 cm or 6 cm will be used, depending on which muscle is visualized in accordance with our routine clinical protocols. During the dynamic approach, the transducer will be placed in a longitudinal fixed position on the muscle using a ProbeFix. All measured contractions in the different muscles will be recorded as short ultrasound videos.
Diagnostic Test: MRI scan — In Stage II, all patients and 10 healthy participants will undergo MRI. During the MRI procedure, we evaluate muscle fat fraction, muscle contractile volume, muscle inflammation and edema.

SUMMARY:
Facioscapulohumeral dystrophy (FSHD) is one of the most common hereditary neuromuscular disorders (NMD), with an estimated prevalence of 2000 patients in the Netherlands. Magnetic resonance imaging (MRI) and muscle ultrasound have contributed to an enhanced understanding of the pathophysiology of Facioscapulohumeral Muscular Dystrophy (FSHD). Previously, our group demonstrated the potential presence of an intermediate factor between muscle fiber loss and clinical weakness in FSHD. The influence of disrupted muscle architecture in FSHD on muscle contractile efficiency is a likely candidate for this factor, and remains relatively unexplored. In this study, we aim to assess the use of ultrasound-defined contractile performance, in comparison with current measures including structural MRI, for monitoring disease progression in FSHD.

DETAILED DESCRIPTION:
Rationale: Facioscapulohumeral dystrophy (FSHD) is a slowly progressive hereditary muscle dystrophy characterized by initial asymmetrical weakness of the facial and shoulder girdle muscles, frequently followed by weakness in the trunk and leg muscles.

Previously, our research group showed the potential presence of an intermediate factor between muscle fiber loss and clinical weakness in FSHD. The influence of disrupted muscle architecture in FSHD on muscle contractile efficiency is a likely candidate for this factor. However, there is currently still a lack of studies on how the disrupted muscle architecture in muscle dystrophies influences the contractile efficiency. We might establish a baseline for muscle contractile performance with muscle ultrasound, determined by muscle strain and displacement.

Muscle imaging has previously contributed to a better understanding of the pathophysiology of various neuromuscular disorders. Both MRI and ultrasound have proven their clinical relevance in neuromuscular dystrophy. With the current development of FSHD clinical trials, the extensive need for biomarkers to follow disease progression is growing. To investigate whether muscle contractile performance can help explain the loss in strength and thereby also has the potential to act as a future biomarker, will be explored in this project.

Objective(s): We aim to assess the use of ultrasound-defined contractile performance as a biomarker for monitoring disease progression and treatment effects in patients with FSHD.

Stage I:

To establish the feasibility, optimal protocol, and repeatability of quantifying ultrasound-defined muscle contractile performance in the upper and lower limb muscles in healthy volunteers and patients with FSHD.

Stage II:

1. To determine the differences in ultrasound-defined contractile performance between healthy individuals and patients with FSHD, and compare to conventional clinical measures, ultrasound measures and MRI measures.
2. To determine the responsiveness of ultrasound-defined contractile performance to disease progression in FSHD patients after 1 year, and compare to MRI measures and other ultrasound measures.

Study design: This prospective cohort study consists of two different stages. In Stage I, the feasibility and repeatability of quantifying ultrasound-defined muscle contractile performance will be assessed in 15 healthy volunteers and 10 patients with FSHD type 1 or 2. Each participant in stage I has to visit the hospital only once. In Stage II, the ultrasound-defined contractile performance, and other ultrasound and MRI outcome measures of healthy volunteers and FSHD patients (type 1 or 2) are compared. In addition, the responsiveness of the different measurements to disease progression after 1 year will be analyzed only in FSHD patients. 50 patients with FSHD will perform these measurements of stage II during the two scheduled visits at baseline (T0) and the two scheduled visits 1-year after the first visit. In stage II, 25 Healthy volunteers will be recruited and will undergo the muscle ultrasound assessment. Only 10 out of 25 healthy volunteers will also undergo the MRI measurements. None of the healthy volunteers will perform follow-up measurements after 1 year. Therefore, 15 healthy volunteers will perform the ultrasound assessment of stage II during 1 visit and 10 healthy volunteers will perform ultrasound measurements during visit 1 and MRI measurements during visit 2 at baseline. A total of 100 individuals will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years.
* Informed consent is given by the participant.
* Ability to read and understand written and spoken instruction in Dutch.
* Willingness and ability to understand nature and content of the study

Exclusion Criteria:

* BMI ≥ 35
* Other diseases that could diffusely affect muscle integrity or disturb the imaging appearance beyond that what can be extrapolated.
* Wheelchair dependence
* Pregnancy
* Stage II: Any contra-indications for MRI, including:

  * Claustrophobia
  * Pacemakers and defibrillators
  * Nerve stimulators
  * Intracranial clips
  * Intraorbital or intraocular metallic fragments
  * Cochlear implants and ferromagnetic implants (e.g. implant for scoliosis)
  * Inability to lie supine for 60 minutes
  * Necessity of (continuous) daytime ventilation
  * Scoliosis surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In the Netherlands, FSHD has an estimated prevalence of 2000 patients. All patients will be recruited from one of the largest longitudinal follow up database, FSHD-FOCUS, which is maintained at the Dutch Radboudumc expertise center. This FSHD-FOCUS cohortwas started in 2014 and includes around 200 patients with clinically and genetically proven FSHD type 1 and type 2. A 5-year-follow-up study (FSHD-FOCUS2) collected comprehensive data on the natural course of FSHD using multiple clinical outcome measures. Only patients who have given consent during the FSHD-FOCUS study to be contacted for subsequent research, will be contacted for this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Stage I: Repeatability and feasibility of the ultrasound-defined muscle contractile performance. | At baseline
  The feasibility of the ultrasound-defined contractile performance procedure is expressed in the number of dropouts in stage I. The repeatability of the muscle contractile performance procedure will be determined with the coefficient of variation in stage I.
Stage II: Difference in contractile performance, MRI measures and clinical measures between healthy individuals and patients with FSHD. | At baseline
  The ultrasound Speckle-Tracking technique is employed during the dynamic approach to establish the muscle contractile performance, determined by muscle strain and displacement. The Ultrafast Shear Wave Elastography Imaging technique is used during the static approach to evaluate muscle stiffness, grey values(Z-scores) and muscle pinnation angle.
  With the MRI measurements we evaluate the muscle fat fraction (%), contractile volume(mm^3), muscle edema, muscle inflammation, fiber curvature, fascicle length(mm), PCSA(mm^2).
Stage II: Change of contractile performance, MRI measures and clinical measures with FSHD disease progression after 1 year. | change from baseline to 1 year follow-up
  The ultrasound, MRI and clinical measures at baseline are compared with the measures after 1 year.
  The ultrasound Speckle-Tracking technique is employed during the dynamic approach to establish the muscle contractile performance, determined by muscle strain and displacement. The Ultrafast Shear Wave Elastography Imaging technique is used during the static approach to evaluate muscle stiffness, grey values(Z-scores) and muscle pinnation angle.
  For FSHD patients in this study the Medical Research Counsel scale (MRC) and/or Ricci score will be known. These measures will also be used to evaluate disease progression. The range of the MRC score is 0-5, in which '0' means no contraction of the muscle and '5' means normal contraction of the muscle. The Ricci score ranges from 0 - 10 (0= no symptoms and 10=wheelchair bound).
  With the MRI measurements we evaluate the muscle fat fraction (%), contractile volume(mm^3), fiber curvature, fascicle length(mm), PCSA(mm^2).

CONTACTS AND LOCATIONS:
Overall Officials: Nens Van Alfen, MD. PhD., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All anonymized (imaging) data will be made available in a suitable open-source online repository after the study results are published in peer-reviewed journals. A DOI will be assigned to dataset published in the Donders Data Repository (soon: Radboud Data Repository).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available after publication for long-term. To guarantee the long-term accessibility of data files, the repository may perform data migration. Even if data is removed, audit trails of 'removed' collections are always retained. Likewise, the metadata of published or archived collections are never removed.
Access Criteria: The data Donders Repository will be used to guarantee long-term accessibility of the research data from this project. The pseudonymized data will be accessible in Donders Repository (soon: Radboud repository (RDR)) under restricted access. Requests for access will be checked, against the conditions for sharing the data as described in the signed Informed Consent. This repository is classified as a highest security-grade data system suitable for preserving large volume, privacy sensitive (i.e. human) research data.
URL: https://data.ru.nl/?10